CLINICAL TRIAL: NCT03261687
Title: The Effects of a Water Based Exercise Programme and a Land Based Exercise Programme on Women Experiencing Pregnancy Related Pelvic Girdle Pain : a Randomised Controlled Feasibility Study.
Brief Title: The Effects of a Water Based Exercise Programme and a Land Based Exercise Programme on Women Experiencing Pregnancy Related Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bradford (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 198588
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy Related; Pelvic Girdle Pain
Keywords: pregnancy; pelvic girdle pain; hydrotherapy; quality of life; physical therapy
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: a randomised controlled feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Exercise + advice (Experimental): Each group undertook four, once weekly exercise sessions (including a warm up, cool down, relaxation, pelvic control and stability exercise). Both programmes focused on similar exercise and muscle groups, but due to the aquatic medium programmes were unable to be exactly matched.
  Interventions: Other: water based exercise; Behavioral: advice
- Land Exercise + advice (Experimental): Each group undertook four, once weekly exercise sessions (including a warm up, cool down, relaxation, pelvic control and stability exercise). Both programmes focused on similar exercise and muscle groups, but due to the aquatic medium programmes were unable to be exactly matched.
  Interventions: Other: land based exercise; Behavioral: advice

INTERVENTIONS:
Other: water based exercise
  Arms: Water Exercise + advice
Other: land based exercise
  Arms: Land Exercise + advice
Behavioral: advice — general advice given to all subjects

SUMMARY:
This study aimed to address whether a water exercise programme improves pain and quality of life in pregnant patients with Pelvic Girdle Pain (PGP) compared to a land-based exercise programme and the feasibility of undertaking a large-scale research programme.

DETAILED DESCRIPTION:
This study aimed to address whether a water exercise programme improves pain and quality of life in pregnant patients with Pelvic Girdle Pain (PGP) compared to a land-based exercise programme and the feasibility of undertaking a large-scale research programme. Twenty-three participants with diagnosed PGP, recruited at St George's Hospital London, were randomised into two groups (water or land exercise). Each group received, four, once-weekly exercise sessions on land or water. Exercise effects on PGP were measured using a variety of outcome measures. Outcomes were assessed at baseline and post four weeks exercise.

ELIGIBILITY:
Inclusion Criteria:

Participants were over eighteen years old, over twelve weeks pregnant and able to speak English.

Exclusion Criteria:

Participants were excluded from the study if they had uncontrolled blood pressure, placenta praevia, pre-eclampsia, obstetric cholestatsis, uncontrolled asthma, unstable respiratory or cardiac conditions, had open skin wounds or MRSA

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Pelvic Girdle Pain Questionnaire (PGPQ) | 4 weeks (pre and post intervention)
  A score change of 7 was set as a clinically significant difference

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 4 weeks (pre and post intervention)
  score change of 1.5 was set as clinically significant
Patient Specific Functional Score (PSFS) | 4 weeks (pre and post intervention)
  score change of 1 was set as clinically significant
Active Straight Leg Raise (ASLR). | 4 weeks (pre and post intervention)
  score change of 1 was set as clinically significant

CONTACTS AND LOCATIONS:
Locations (1):
- St George's Hospital,, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No